CLINICAL TRIAL: NCT04535947
Title: A Phase 2, Multicenter, Double-Masked, Randomized, Vehicle-Controlled, Parallel Group, Study of SDP-4 Ophthalmic Solution in Subjects With Dry Eye Disease (DED)
Brief Title: Study to Evaluate the Efficacy of SDP-4 in Subjects With Dry Eye Disease (DED) (SDP-4-CS202)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Silk Technologies, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SDP-4-CS202
Record Dates: First submitted 2020-08-27; First posted 2020-09-02 (Actual); Results first posted 2022-09-01 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2021-05

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to either 1% SDP-4 ophthalmic solution or vehicle in 1:1 ratio in parallel groups.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All investigation product (1% SDP-4 ophthalmic solution and vehicle) will be provided in single-use doses (SUDs) contained in foil pouches.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vehicle (Placebo Comparator): Vehicle
  Interventions: Drug: Vehicle
- SDP-4 Ophthalmic Solution (1.0%) (Experimental): Active
  Interventions: Drug: SDP-4 Ophthalmic Solution (1.0%)

INTERVENTIONS:
Drug: Vehicle — Investigational product (IP) will be administered via topical ocular instillation, one drop per eye, twice daily (BID) for 8 weeks (56 days). Both eyes will be treated.
  Arms: Vehicle
Drug: SDP-4 Ophthalmic Solution (1.0%) — Investigational product (IP) will be administered via topical ocular instillation, one drop per eye, twice daily (BID) for 8 weeks (56 days). Both eyes will be treated.
  Other Names: SDP-4 (1.0%)
  Arms: SDP-4 Ophthalmic Solution (1.0%)

SUMMARY:
SDP-4-CS202 is a Phase 2, multicenter, double-masked, randomized, vehicle-controlled, parallel group study designed to evaluate the ocular efficacy of SDP-4 ophthalmic solution in subjects with moderate to severe dry eye disease over an 8-week treatment period. Once concentration (1%) of SDP-4 ophthalmic solution will be given in a parallel group to vehicle via topical ocular instillation BID.

ELIGIBILITY:
Inclusion Criteria:

* Have DED in both eyes, as supported by a subject-reported history of daily symptoms of dryeye for ≥ 6 months prior to Visit 1/Screening requiring the use of artificial tears.
* Total score ≥ 40 and ≤ 70 on the SANDE questionnaire at Visits 1 and 2.
* Tear break-up time (TBUT) of ≤ 6 seconds in both eyes at Visits 1 and 2.
* Anesthetized Schirmer's test tear volume ≥ 3 mm and <10 mm in both eyes (only at Visit 1).
* Best-corrected visual acuity (BCVA) of +0.7 logMAR or better in each eye as assessed by logMAR chart at Visits 1 and 2.

Exclusion Criteria:

* Ocular surface corneal disease other than DED.
* Diagnosis of Sjögren's disease.
* Lid margin disorder other than meibomian gland dysfunction (MGD)
* Presence of any ocular condition (e.g., pterygium) that in the Investigator's opinion could affect study parameters.
* Any previous reconstructive or cosmetic eyelid surgery
* Any previous invasive glaucoma and/or corneal surgery
* Corneal refractive surgery in the 12 months prior to Visit 1/Screening.
* Cataract extraction within 90 days prior to Visit 1/Screening.
* Cauterization of the punctum or punctal plug (silicone or collagen) insertion or removal within 30 days prior to Visit 1/Screening or planned during the study.
* Contact lens wear.
* Use of ophthlamic corticosteroids, NSAIDs, antibiotics, antihistamines, IOP lowering medication, in the 30 days prior to Visit 1/Screening
* Serious systemic disease or uncontrolled medical condition that in the judgment of the Investigator could confound study assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2020-08-14 (Actual); Primary Completion 2021-02-10 (Actual); Study Completion 2021-02-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Orange County Ophthalmology Medical Group, Garden Grove, California
  - LoBue Laser and Eye Medical Center, Murrieta, California
  - Eye Research Foundation, Newport Beach, California
  - Ophthalmology Associates, St Louis, Missouri
  - Total Eye Care, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vehicle | SDP-4 Ophthalmic Solution (1.0%)
Started | 76 | 77
Completed | 72 | 72
Not Completed | 4 | 5
Not completed — Adverse Event | 1 | 4
Not completed — Other reasons not specified | 2 | 0
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vehicle | SDP-4 Ophthalmic Solution (1.0%) | Total
Number analyzed (Participants) | 76 | 77 | 153
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (15.18) | 58.8 (14.95) | 60.2 (15.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 55 | 107
  Male | 24 | 22 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 14 | 23
  Not Hispanic or Latino | 67 | 63 | 130
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 13 | 12 | 25
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 8 | 10 | 18
  White | 54 | 54 | 108
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Iris Color [Count of Participants; unit: Participants]
  Blue | 20 | 11 | 31
  Brown | 42 | 45 | 87
  Green | 3 | 6 | 9
  Hazel | 11 | 15 | 26

OUTCOME MEASURES:

1. Primary Outcome: Symptom Assessment in Dry Eye (SANDE) Questionnaire
Description: Mean change from baseline in total SANDE at Visit 5/Day 56
  The SANDE questionnaire contained two questions regarding the frequency and severity of DED symptoms, with a total score being the square root of the frequency score times the square root of the severity score (range 0 100). A higher score indicates more severe DED symptoms.
Time Frame: 56 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vehicle | SDP-4 Ophthalmic Solution (1.0%)
Number analyzed (Participants) | 72 | 72
units on a scale
  Screening | 58.95 (6.635) | 57.21 (7.850)
  Day 56 | -18.80 (22.288) | -16.60 (19.075)

2. Secondary Outcome: Corneal Fluorescein Staining
Description: Mean and mean change from baseline at each visit
  Reported on a scale of 0-15 with values greater than 3 indicating abnormal incidence of corneal surface irregularity.
Time Frame: 56 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vehicle | SDP-4 Ophthalmic Solution (1.0%)
Number analyzed (Participants) | 72 | 72
units on a scale
  Screening | 0.68 (0.697) | 0.74 (0.696)
  Day 14 | -0.21 (0.664) | -0.04 (0.772)
  Day 28 | -0.15 (0.660) | -0.22 (0.809)
  Day 56 | -0.15 (0.725) | -0.24 (0.682)

3. Secondary Outcome: Tear Breakup Time
Description: Mean and mean change from baseline at each visit
Time Frame: 56 days
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Vehicle | SDP-4 Ophthalmic Solution (1.0%)
Number analyzed (Participants) | 72 | 72
seconds
  Day 1 | 3.75 (1.104) | 3.80 (0.990)
  Day 14 | 1.06 (2.570) | 1.42 (2.850)
  Day 28 | 2.00 (2.596) | 1.95 (4.069)
  Day 56 | 1.77 (2.865) | 1.80 (2.419)

4. Secondary Outcome: Conjunctival Hyperemia
Description: Mean and mean change from baseline at each visit
  Reported on a scale of 0-15 with values greater than 3 indicating abnormal incidence of conjunctival surface irregularity.
Time Frame: 56 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vehicle | SDP-4 Ophthalmic Solution (1.0%)
Number analyzed (Participants) | 72 | 72
units on a scale
  Day 1 Baseline | 0.80 (0.833) | 0.91 (0.948)
  Day 14 | 0.00 (0.520) | 0.01 (0.425)
  Day 28 | -0.07 (0.608) | -0.03 (0.530)
  Day 56 | 0.03 (0.604) | -0.06 (0.554)

5. Secondary Outcome: Individual Symptom Visual Analog Scale (VAS) Scores, Separately for Each Symptom (Burning / Stinging)
Description: Mean and mean change from baseline at final visit as measured on a scale from 0 to 100, where higher scores indicate a worse outcome
Time Frame: 56 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vehicle | SDP-4 Ophthalmic Solution (1.0%)
Number analyzed (Participants) | 72 | 72
units on a scale | -7.89 (22.985) | -17.06 (23.356)

6. Secondary Outcome: Individual Symptom Visual Analog Scale (VAS) Scores, Separately for Each Symptom (Eye Discomfort)
Description: as for outcome 5
Time Frame: 56 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vehicle | SDP-4 Ophthalmic Solution (1.0%)
Number analyzed (Participants) | 72 | 72
units on a scale | -12.10 (21.195) | -13.18 (22.283)

7. Secondary Outcome: Individual Symptom Visual Analog Scale (VAS) Scores, Separately for Each Symptom (Eye Dryness)
Description: as for outcome 5
Time Frame: 56 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vehicle | SDP-4 Ophthalmic Solution (1.0%)
Number analyzed (Participants) | 72 | 72
units on a scale | -17.97 (24.768) | -18.38 (20.921)

8. Secondary Outcome: Individual Symptom Visual Analog Scale (VAS) Scores, Separately for Each Symptom (Eye Pain)
Description: as for outcome 5
Time Frame: 56 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vehicle | SDP-4 Ophthalmic Solution (1.0%)
Number analyzed (Participants) | 72 | 72
units on a scale | -6.94 (21.200) | -6.47 (23.400)

9. Secondary Outcome: Individual Symptom Visual Analog Scale (VAS) Scores, Separately for Each Symptom (Fluctuating Vision)
Description: as for outcome 5
Time Frame: 56 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vehicle | SDP-4 Ophthalmic Solution (1.0%)
Number analyzed (Participants) | 72 | 72
units on a scale | -6.17 (20.025) | -8.11 (20.654)

10. Secondary Outcome: Individual Symptom Visual Analog Scale (VAS) Scores, Separately for Each Symptom (Foreign Body Sensation)
Description: as for outcome 5
Time Frame: 56 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vehicle | SDP-4 Ophthalmic Solution (1.0%)
Number analyzed (Participants) | 72 | 72
units on a scale | -6.94 (20.567) | -10.58 (20.031)

11. Secondary Outcome: Individual Symptom Visual Analog Scale (VAS) Scores, Separately for Each Symptom (Itching)
Description: as for outcome 5
Time Frame: 56 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vehicle | SDP-4 Ophthalmic Solution (1.0%)
Number analyzed (Participants) | 72 | 72
units on a scale | -13.81 (24.411) | -9.75 (22.890)

12. Secondary Outcome: Individual Symptom Visual Analog Scale (VAS) Scores, Separately for Each Symptom (Photophobia)
Description: as for outcome 5
Time Frame: 56 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vehicle | SDP-4 Ophthalmic Solution (1.0%)
Number analyzed (Participants) | 72 | 72
units on a scale | -12.69 (21.512) | -10.43 (22.143)

ADVERSE EVENTS:
Time Frame: 56 days
Arm/Group | Vehicle | SDP-4 Ophthalmic Solution (1.0%)
All-Cause Mortality (participants affected / at risk) | 0/76 | 0/77
Serious Adverse Events (participants affected / at risk) | 0/76 | 1/77
Other Adverse Events (participants affected / at risk) | 8/76 | 8/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vehicle (N=76) | SDP-4 Ophthalmic Solution (1.0%) (N=77)
Detached Retina (Eye disorders) | 0 (0) | 1 (1) — One subject reported recent loss of vision, was diagnosed with a macula off retinal detachment with blurred vision during the course of the study. The event was judged not related to SDP-4 treatment.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vehicle (N=76) | SDP-4 Ophthalmic Solution (1.0%) (N=77)
Eye Pain (Eye disorders) | 0 (0) | 1 (1)
Installation Site Pain (General disorders) | 5 (10) | 4 (8)
Blepharitis (Eye disorders) | 1 (2) | 1 (1)
Conjunctivitis Allergic (Eye disorders) | 0 (0) | 1 (2)
Cystoid macular oedema (Eye disorders) | 0 (0) | 1 (1)
Eyelid Oedema (Eye disorders) | 0 (0) | 1 (1)
Eyelid Ptosis (Eye disorders) | 0 (0) | 1 (1)
Retinal Detachment (Eye disorders) | 0 (0) | 1 (1)
Vision Blurred (Eye disorders) | 0 (0) | 1 (1)
Visual Acuity Reduced (Eye disorders) | 0 (0) | 1 (1)
Installation Site Discomfort (General disorders) | 2 (4) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All information concerning SDP-4 and the operations of Silk Technologies, such as patent applications, formulas, manufacturing processes, basic scientific data or formulation information not previously published, are considered CONFIDENTIAL and shall remain the sole property of Silk Technologies. The Investigator agrees to use this information only in accomplishing this study and will not use it for other purposes without the written consent of Silk Technologies

DOCUMENTS (3):
  • Study Protocol (2020-03-12): https://cdn.clinicaltrials.gov/large-docs/47/NCT04535947/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-24): https://cdn.clinicaltrials.gov/large-docs/47/NCT04535947/SAP_001.pdf
  • Informed Consent Form (2020-03-16): https://cdn.clinicaltrials.gov/large-docs/47/NCT04535947/ICF_002.pdf